CLINICAL TRIAL: NCT05479331
Title: The Relationship Between Sarcopenia and Cardiovascular Disease in Chronic Kidney Disease Stage 3 or Higher and the Risk Involved.
Brief Title: The Relationship Between Sarcopenia and Cardiovascular Disease in Chronic Kidney Disease and the Risk Involved.
Status: Completed | Type: Observational
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Na Jiang, Associate Chief Physician of Nephrology, Shanghai Jiao Tong University School of Medicine
Other Study IDs: sarcopenia
Record Dates: First submitted 2022-07-27; First posted 2022-07-29 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2019-12

CONDITIONS: Sarcopenia; CKD; Cardiovascular Diseases
MeSH Terms: conditions — Sarcopenia; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- sarcopenia: CKD patients with sarcopenia, meeting the following two criteria (1) male LTI (lean tissue index)< 7.0 kg/m2, female LTI < 5.7 kg/m2; (2) Male HGS)(handgrip strength < 26 kg, female HGS < 18 kg.
- non-sarcopenia: CKD patients with non-sarcopenia

SUMMARY:
This study explores the risk factors for sarcopenia in patients with chronic kidney disease and the effects of sarcopenia on cardiovascular disease. Treatment of sarcopenia and cardiovascular complications provides a basis for improving the quality of life and survival of patients with chronic kidney disease.

DETAILED DESCRIPTION:
Sarcopeniais a syndrome characterized by the loss of skeletal muscle mass, muscle strength, and muscle dysfunction. The high incidence of sarcopenia in patients with chronic kidney disease (CKD) is strongly associated with poor quality of life, cardiovascular events, and increased all-cause mortality. At present, the cause of sarcopenia in patients with CKD is still unclear, and factors such as inflammation, malnutrition, and hormone metabolism disorders may affect the occurrence and development of sarcopenia. This topic explores the risk factors of sarcopenia in patients with chronic kidney disease and the correlation between sarcopenia and the risk of cardiovascular disease, and provides a basis for the prevention and treatment of sarcopenia and cardiovascular complications, with a view to improving the prognosis of CKD patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients presented by the Nephrology Center during August 2019 and March 2021
* Age 18-75 years;
* Patients with CKD2 or above (eGFR≤60 ml/(min 1.73m2)

Exclusion Criteria:

* There are contraindications to bioelectrical impedance spectroscopy (BIS) . examination, such as amputation, metal implants in the body, etc.;
* Complicated with other serious diseases, such as malignant tumors, cirrhosis, systemic infections, etc.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with chronic kidney disease
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Epicardial adipose tissue measured by ultrasound color doppler | the day when being recruited
  EAT is defined as a fat depot that exists on the surface of the myocardium,which plays a detrimental role in our health. EAT would be measured by ultrasound color doppler.
Intima-media thickness measured by ultrasound color doppler | the day when being recruited
  IMT of carotid arteries, as assessed noninvasively by carotid ultrasonography, is a useful measure of preclinical atherosclerosis. Carotid IMT has been found to predict future risk of cardiovascular disease.IMT would be measured by ultrasound color doppler.

SECONDARY OUTCOMES:
Baseline demographic, clinical and laboratory characteristics | the day when being recruited
  Demographic characteristics include age, sex, height, body mass, blood pressure, primary disease, and comorbidities. BMI = the square of body weight/height (kg/m2). Patient comorbidities were assessed using the Charlson comorbidity Index (CCI). Subjective global assessment (SGA) was used to assess the nutritional status of patients. Laboratory characteristics include sALB,Pre-alb,hs-CRP,TC,TAG,LDL-C,HDL-C,PG ,HbA1c ,creatinine,BNP,iPTH,etc.

CONTACTS AND LOCATIONS:
Overall Officials: Jiangzi Yuan, MD, Study Director — Baoshan Site of Ren Ji Hospital, School of Medicine, Shanghai Jiaotong University
Locations (1):
- Baoshan Site of Shanghai Renji Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No